CLINICAL TRIAL: NCT04411784
Title: PROTECT-ASUC: Covid-19 Pandemic Response Of assessmenT, EndosCopy and Treatment in Acute Severe Ulcerative Colitis: A Multi-centre Observational Case- Control Study
Brief Title: PROTECT-ASUC: Covid-19 Pandemic Response Of assessmenT, EndosCopy and Treatment in Acute Severe Ulcerative Colitis
Acronym: PROTECT-ASUC
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 284030
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Inflammatory Bowel Diseases; COVID
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main group: Patient with Acute Severe Ulcerative Colitis based on Modified Truelove and Witts Severity Index managed during the study period
- Control Group: Patients with ASUC managed in the unit from 1st Jan to 31st June 2019

SUMMARY:
Whether the perceived changes in management of Acute Severe Ulcerative Colitis during the COVID pandemic are widespread, and whether they have any impact on patient outcomes

DETAILED DESCRIPTION:
The study aims to evaluate the process, evaluation and therapy variation in management of ASUC with reference to 2019 British Society of Gastroenterology guidelines and see whether there are any differences between ambulatory and hospital management in ASUC. Also to evaluate the outcomes in ASUC patients managed during the COVID-19 pandemic

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 -100 inclusive
* Acute Severe Ulcerative Colitis based on Modified Truelove and Witts Severity Index managed during the study period

Exclusion Criteria:

* Patients aged 16 -100 inclusive
* Acute Severe Ulcerative Colitis based on Modified Truelove and Witts Severity Index managed during the study period

  * Admission for elective colectomy
  * Pouch or stoma

Ages: 16 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In The UK alone approximately 6500 patients are admitted with ASUC each year
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure: The need for in-hospital colectomy or rescue therapy | 3 months
  The need for in-hospital colectomy or rescue therapy

SECONDARY OUTCOMES:
2.1: Duration and type/route of steroid use | 3 months
  Duration and type/route of steroid use
2.2: 30 day colectomy free survival rates | 3 months
  30 day colectomy free survival rates
2.3: Covid-19 infection rates | 3 months
  Covid-19 infection rates
2.4: Rate of Rescue therapy use | 3 months
  Rate of Rescue therapy use
2.5: Duration of hospital stay | 3 months
  Duration of hospital stay
2.6: Admission severity scoring | 3 months
  Admission severity scoring
2.7: Readmission rates | 3 months
  Readmission rates

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Sebastian, Principal Investigator — Hull University Teaching Hospitals
Locations (1):
- Gastroenterology, Hull Royal Infirmary, Hull University Teaaching Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sebastian S, Patel KV, Segal JP, Subramanian S, Conley TE, Gonzalez HA, Kent AJ, Saifuddin A, Hicks L, Mehta S, Bhala N, Brookes MJ, Lamb CA, Kennedy NA; PROTECT ASUC collaborators; Walker GJ. Ambulatory care management of 69 patients with acute severe ulcerative colitis in comparison to 695 inpatients: insights from a multicentre UK cohort study. BMJ Open Gastroenterol. 2022 Jan;9(1):e000763. doi: 10.1136/bmjgast-2021-000763. PMID 35101886
- [Derived] Sebastian S, Walker GJ, Kennedy NA, Conley TE, Patel KV, Subramanian S, Kent AJ, Segal JP, Brookes MJ, Bhala N, Gonzalez HA, Hicks LC, Mehta SJ, Lamb CA; PROTECT-ASUC Study Group. Assessment, endoscopy, and treatment in patients with acute severe ulcerative colitis during the COVID-19 pandemic (PROTECT-ASUC): a multicentre, observational, case-control study. Lancet Gastroenterol Hepatol. 2021 Apr;6(4):271-281. doi: 10.1016/S2468-1253(21)00016-9. Epub 2021 Feb 2. PMID 33545083